CLINICAL TRIAL: NCT04370028
Title: All-Russian Observational Non-interventional Study on Efficacy and Safety of Divaza in Patients With Chronic Cerebral Ischemia and Cognitive Disorders
Brief Title: Study on Efficacy and Safety of Divaza in Patients With Chronic Cerebral Ischemia and Cognitive Disorders
Acronym: DIAMANT
Status: Completed | Type: Observational
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Other Study IDs: DIAMANT
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-04

CONDITIONS: Chronic Cerebral Ischemia
MeSH Terms: interventions — divaza

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Divaza: Oral administration. 2 tablet 3 times daily. Keep the tablets in the mouth until completely dissolved, outside of meal.
  Interventions: Drug: Divaza

INTERVENTIONS:
Drug: Divaza — Oral administration.

SUMMARY:
An open-label, prospective, observational, multicenter study. The study enrolls adult outpatients with CCI from 8 federal districts of the Russian Federation.

DETAILED DESCRIPTION:
Medical data (demographic and clinical characteristics - diagnosis, MoCA test results) are collected from patients to whom Divaza is prescribed to be taken according to the following regimen: 2 tablets 3 times per day for 12 weeks.

Neurologists assess the patients' cognitive functions with MoCA scale before starting therapy with Divaza (visit 1) and 12 weeks after the treatment (visit 2).

The efficacy of Divaza for the treatment of cognitive impairment in patients with chronic cerebral ischemia (CCI) is evaluated.

Safety is assessed based on the frequency and severity of adverse events. In addition, the relationship between MoCA test performance and gender or regional social and economic factors is evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender aged 18+ years.
2. Diagnosis of chronic cerebral ischemia (CCI) based on the clinical history of underlying vascular disease(atherosclerosis and/or arterial hypertension) and neurological signs.
3. Unchanged basic therapy of CCI and underlying vascular disease for a previous 3 month.
4. Signed informed consent form.

Exclusion Criteria:

1. Other neurological diseases.
2. Any known allergy to/intolerance of any constituent of the medication.
3. Pregnancy, breast-feeding.
4. Participation in other clinical trials for 3 months prior to enrollment in this study.
5. The patient is related to the research personnel of the investigative sites that are directly involved in the study, or is the immediate relative of the investigator, or the employee of OOO NPF Materia Medica Holding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CCI outpatients with cognitive impairment (MoCA score <26) or without one (MoCA score ≥ 26) recieving unchanged basic therapy of CCI and underlying vascular disease for a 3 month previous to the onset of the study. Diagnosis of сhronic cerebral ischemia (CCI) was based on the clinical history of underlying vascular disease(atherosclerosis and/or arterial hypertension) and neurological signs. Vascular nature of cognitive impairment in patients with MoCA<26 was determined according to NINDS-AIREN criteria.
Sampling Method: Probability Sample
Enrollment: 2583 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 2016 January 2017 Location: outpatient clinics from 8 federal districts of the Russian Federation
Groups:
- Divaza Treatment Group: All enrolled patients received Divaza 2 tablets 3 times per day for 12 weeks
Period: Overall Study
Arm/Group | Divaza Treatment Group
Started | 2583
Completed | 1876
Not Completed | 707
Not completed — Withdrawal by Subject | 695
Not completed — Protocol Violation | 9
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Safety was assessed using the data of all 2583 patients. Within each efficacy and demographic analysis only complete cases approach was used, therefore the number of patients analyzed in efficacy analysis was fewer than 1876
Groups:
- Divaza Treatment Group: All participants received Divaza treatment
Arm/Group | Divaza Treatment Group
Number analyzed (Participants) | 1876
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not reported for 23 patients.
  years
    number analyzed (Participants) | 1853
    (all) | 65.7 (19.1)
Age, Customized [Number; unit: participants] — Population: Age was not reported for 23 patients
  participants
    Young (<35 yo): number analyzed (Participants) | 1853
    Young (<35 yo) | 25
    Middle aged (35-59 yo): number analyzed (Participants) | 1853
    Middle aged (35-59 yo) | 501
    Elderly (60-75 yo): number analyzed (Participants) | 1853
    Elderly (60-75 yo) | 1062
    Senile (75-90 yo): number analyzed (Participants) | 1853
    Senile (75-90 yo) | 265
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Within each analysis only complete cases approach was used.Sexual identity of 29 patients was not specified.
  Participants
    number analyzed (Participants) | 1847
    Female | 1139
    Male | 708
Baseline MoCA score [Mean (Standard Deviation); unit: units on a scale] — MoCA - Montreal Cognitive Assessment (0-30 scores, higher scores mean a better outcome).MoCA test allows to evaluate the presence of cognitive impairment Population: Baseline MoCA scores were not reported in 21 patients.
  units on a scale
    number analyzed (Participants) | 1855
    (all) | 19.4 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean MoCA Score at Week 1 and the End of the 12-week Therapy
Description: MoCA - Montreal Cognitive Assessment (0-30 scores, higher scores mean a better outcome).MoCA test allows to evaluate the presence of cognitive impairment
Time Frame: week 1 to 12 week
Population: MoCA scores were not reported in 21 patients at least at one timepoint (excluded from analysis)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Divaza Treatment Group: All analyzed participants received Divaza treatment 2 tablets 3 times per day for 12 weeks
Arm/Group | Divaza Treatment Group
Number analyzed (Participants) | 1855
score on a scale
  1 week | 19.42 (5.13)
  12 week | 24 (4.6)
Statistical Analysis 1: Comparison: Divaza Treatment Group; Test type: Superiority; p < 0.00001, t-test, 2 sided; Paired test was performed; Mean Difference (Net) = 4.57, 95% CI 2-sided [4.42 to 4.72]

2. Secondary Outcome: The Number of Patients With a MoCA Score <26 at 12 Week
Description: The number of patients with mild cognitive impairment. MoCA - Montreal Cognitive Assessment (0-30 scores, higher scores mean a better outcome)
Time Frame: 12 week
Population: MoCA scores were not reported in 21 patients at least at one timepoint (excluded from analysis)
Measure: Number; unit: participants
Arm/Group | Divaza Treatment Group
Number analyzed (Participants) | 1855
participants
  week 1 | 1676
  week 12 | 1048
Statistical Analysis 1: Comparison: Divaza Treatment Group; Odds ratio of occuring MoCA score <26 was assessed; Test type: Superiority; p < 0.00001, Fisher Exact; Odds Ratio (OR) = 7.2, 95% CI 2-sided [6.01 to 8.67] — OR estimated (week 1 to week 12) the higher the better

3. Secondary Outcome: The Number of Patients With a MoCA Score ≤ 17 at the End of the 12-week Therapy
Description: The number of patients with dementia. MoCA - Montreal Cognitive Assessment (0-30 scores, higher scores mean a better outcome)
Time Frame: week1 to week 12
Population: MoCA scores were not reported in 21 patients at least at one timepoint (excluded from analysis)
Measure: Number; unit: participants
Arm/Group | Divaza Treatment Group
Number analyzed (Participants) | 1855
participants
  week 1 | 489
  week 12 | 117
Statistical Analysis 1: Comparison: Divaza Treatment Group; Odds ratio of occuring MoCA score <17 was assessed; Test type: Superiority; p < 0.00001, Fisher Exact; Odds Ratio (OR) = 5.31, 95% CI 2-sided [4.28 to 6.64] — OR estimated (week 1 to week 12) the higher the better

4. Secondary Outcome: The Dynamics of Mean MoCA Score in Each Age Group
Description: Age groups:young <35 yo, middle-aged - 35-59 yo, elderly - 60-75 yo, senile - 75-90 yo MoCA - Montreal Cognitive Assessment (0-30 scores, higher scores mean a better outcome)
Time Frame: week1 to week 12
Population: Patients who did not reported age or both MoCA scores were excluded from analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Young Patients<35 yo: Young Patients<35 yo treated with Divaza
- Middle-aged Patients 35-59 yo: Middle-aged patients 35-59 yo treated with Divaza
- Elderly Patients 60-75 yo: Elderly patients 60-75 yo treated with Divaza
- Senile Patients 75-90 yo: Senile patients 75-90 yo received Divaza
Arm/Group | Young Patients<35 yo | Middle-aged Patients 35-59 yo | Elderly Patients 60-75 yo | Senile Patients 75-90 yo
Number analyzed (Participants) | 25 | 501 | 1062 | 265
score on a scale
  week 1 | 24 (5.6) | 20.94 (4.93) | 19.39 (4.7) | 16.23 (5.42)
  week 12 | 26.4 (5.6) | 25.7 (3.6) | 23.9 (4.2) | 20.7 (5.6)
Statistical Analysis 1: Comparison: Young Patients<35 yo; Change of mean MoCA score; Test type: Superiority; p < 0.07, ANOVA; Mean Difference (Net) = 2.375, 95% CI 2-sided [-0.21 to 4.96]
Statistical Analysis 2: Comparison: Middle-aged Patients 35-59 yo; Change of mean MoCA score; Test type: Superiority; p < 0.01, ANOVA; Mean Difference (Net) = 4.74, 95% CI 2-sided [4.17 to 5.31]
Statistical Analysis 3: Comparison: Elderly Patients 60-75 yo; Change of mean MoCA score; Test type: Superiority; p < 0.01, ANOVA; Mean Difference (Net) = 4.55, 95% CI 2-sided [4.16 to 4.94]
Statistical Analysis 4: Comparison: Senile Patients 75-90 yo; Change of mean MoCA score; Test type: Superiority; p < 0.01, ANOVA; Mean Difference (Net) = 4.49, 95% CI 2-sided [3.7 to 5.27]

5. Secondary Outcome: The Number of Patients With a MoCA Score Improvement (Increase in Scores) in Age Groups
Description: as for outcome 4
Time Frame: week1 to week 12
Population: Patients who did not reported age or both MoCA scores were excluded from analysis
Measure: Number; unit: participants
Arm/Group | Young Patients<35 yo | Middle-aged Patients 35-59 yo | Elderly Patients 60-75 yo | Senile Patients 75-90 yo
Number analyzed (Participants) | 25 | 501 | 1062 | 265
participants | 5 | 199 | 616 | 214

6. Other Pre Specified Outcome: The Relationship Between Cognitive Impairment and Patients' Gender
Description: Evaluation of the relationship between baseline MoCA test results and gender. MoCA - Montreal Cognitive Assessment (0-30 scores, higher scores mean a better outcome)
Time Frame: Data measured at baseline
Population: Patients who did not reported sex or baseline MoCA score were excluded from analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Female: Female patients treated with Divaza
- Male: Male patients treated with Divaza
Arm/Group | Female | Male
Number analyzed (Participants) | 1139 | 708
units on a scale | 19.7 (5.09) | 18.9 (5.13)
Statistical Analysis 1: Comparison: Female vs Male; Test type: Superiority; p = 0.0011, ANOVA; Mean Difference (Net) = 0.803, 95% CI 2-sided [0.321 to 1.28], Standard Error of Mean 0.246

7. Other Pre Specified Outcome: The Relationship Between Cognitive Impairment and Regional Social/Economic Factors
Description: Evaluation of the relationship between baseline MoCA test results and regional developmental social or economic indicators (poverty, infant mortality, migration, life expectancy, innovation rate, professional development, number of university students, number of R&D personnel, resources spent on R&D, number of doctors, number of hospitals and outpatient clinics, hospital capacity, fertility rate, quality of life index,income).
  Relevance of factors (unitless value) provided. The higher the more influential the factor is.
  Relevance was assessed with Boruta approach:
  KURSA, Miron B.; RUDNICKI, Witold R.. Feature Selection with the Boruta Package. Journal of Statistical Software, [S.l.], v. 36, Issue 11, p. 1 - 13, sep. 2010. ISSN 1548-7660. Available at: <http://www.jstatsoft.org/v036/i11>. Date accessed: 24 nov. 2020. doi:http://dx.doi.org/10.18637/jss.v036.i11.
Time Frame: Data measured at baseline
Population: Incomplete data (with respect to used variables) was excluded
Measure: Median (Inter-Quartile Range); unit: unitless feature importance
Arm/Group | Divaza Treatment Group
Number analyzed (Participants) | 1797
unitless feature importance
  Age | 39.85 [39.48 to 41.03]
  Poverty percentage | 8.36 [7.66 to 8.9]
  Infant mortality | 7.97 [7.53 to 8.33]
  Migration index | 7.92 [7.23 to 8.42]
  Life expectancy | 6.42 [5.86 to 7.15]
  Professional development index | 6.13 [5.52 to 6.68]
  Number of R&D personnel | 5.81 [4.7 to 6.37]
  Hospitals number | 5.65 [5.16 to 6.09]
  R&D expenditures | 5.6 [5 to 6.31]
  Innovation rate | 5.56 [5.12 to 6.04]
  Hospitals capacity | 4.89 [4.46 to 5.16]
  Fertility rate | 4.87 [4.3 to 5.41]
  QoL index | 4.85 [4.06 to 5.54]
  Outpatient clinics | 4.73 [4.32 to 5.59]
  Nursing personnel | 4.69 [3.87 to 5.63]
  Income level | 3.83 [3 to 4.59]
  University students | 3.79 [3.19 to 4.33]
  Number of doctors | 3.78 [3.17 to 4.19]
  shadowMax (reference zero-importance feature) | 2.66 [1.83 to 3.11]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: AEs were collected from all patients received a single dose of Divaza according to patient's complaints and physical examination.
Arm/Group | Divaza Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/2583
Serious Adverse Events (participants affected / at risk) | 0/2583
Other Adverse Events (participants affected / at risk) | 17/2583
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Divaza Treatment Group (N=2583)
Nausea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No